CLINICAL TRIAL: NCT03914222
Title: Comparison of Noninvasive Pulmonary Artery Compliance During and After Decompensation in Heart Failure Patients
Brief Title: Comparing PA Compliance During and After Decompensation in HFP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Theranova, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CRD-02-1434
Record Dates: First submitted 2019-04-01; First posted 2019-04-16 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-04

CONDITIONS: Congestive Heart Failure; Decompensated Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- CardioSpire Device (Other): Patients blows into Respirix device or uses BIPAP machine for a few breaths solely to obtain signal.
  Interventions: Device: CardioSpire (Respirix) Device

INTERVENTIONS:
Device: CardioSpire (Respirix) Device — Patients will blow into the device through a small tube, which analyzes the signals in the airway patterns.

SUMMARY:
Pulmonary Artery Compliance measurements will be obtained with the Respirix device in patients with congestive heart failure decompensation. Echocardiogram, weight measurements, and BNP will also be gathered as independent measures of decompensation in the clinic. Pulmonary Artery Compliance measurements will be made daily during the hospital stay. Patients can continue using the device at home for the next 3 weeks. Each patient will serve as their own control and relative changes from their baseline will be recorded for each parameter.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must ≥ 18 years of age
2. Patient has been diagnosed with Congestive Heart Failure, class II-IV
3. Patient is currently being admitted for decompensation related to Congestive Heart Failure
4. Subject or subject's legally authorized representative is able to give informed consent before entering the study.

Exclusion Criteria:

1. Currently pregnant or breastfeeding
2. Clinical signs or symptoms of a respiratory infection
3. Unable to obtain a high-quality signal, as determined by variability of nPAC values throughout a single breath, within 48 hours of enrollment
4. Inability to withstand a 10 second end-inspiratory pause, in the opinion of the investigator
5. Deemed unsuitable for enrollment in study by the investigator based on subjects' history or physical examination

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-06-24 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Diuretics resulting in fluid status changes in severely compensated CHF patients from hospital admit time to discharge and to follow up visit | Through study completion, up to 1 month depending on readmission
  Comparing fluid management (diuretics) to daily CardioSpire's non-invasive Pulmonary Artery Compliance (nPAC) value over the time course from decompensation (at hospital admission) through compensation (discharge) and at their follow up visit, in congestive heart failure patients (CHF).
Vasoactives resulting in fluid status changes in severely compensated CHF patients from hospital admit time to discharge and to follow up visit | Through study completion, up to 1 month depending on readmission
  Comparing fluid management (vasoactives) to daily CardioSpire's non-invasive Pulmonary Artery Compliance (nPAC) value over the time course from decompensation (at hospital admission) through compensation (discharge) and at their follow up visit, in congestive heart failure patients (CHF).
Fluid status based on weight changes in severely compensated CHF patients from hospital admit time to discharge and to follow up visit | Through study completion, up to 1 month depending on readmission
  Comparing fluid management (through weight changes) to daily CardioSpire's non-invasive Pulmonary Artery Compliance (nPAC) value over the time course from decompensation (at hospital admission) through compensation (discharge) and at their follow up visit, in congestive heart failure patients (CHF).
Clinical congestion measurement changes in severely compensated CHF patients from hospital admit time to discharge and to follow up visit | Through study completion, up to 1 month depending on readmission
  Comparing clinical congestion measurement (taken as standard of care) to daily CardioSpire's non-invasive Pulmonary Artery Compliance (nPAC) value over the time course from decompensation (at hospital admission) through compensation (discharge) and at their follow up visit, in congestive heart failure patients (CHF).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Kansas, Kansas City, Kansas, United States